CLINICAL TRIAL: NCT04205032
Title: Evaluation in Healthy Volunteers of CARDIOSPACE II for Physiological Studies in Space
Brief Title: Evaluation in Healthy Volunteers of CARDIOSPACE II
Acronym: CDSII
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Angers (Other Government)
Collaborators: Centre National des Etudes Spatiales - French Space Agency (CNES) (Unknown); Astronautic Center of China (ACC) (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: IRCB:2019-AO1519-48
Record Dates: First submitted 2019-12-11; First posted 2019-12-19 (Actual); Last update posted 2021-07-28 (Actual); Status verified 2021-07

CONDITIONS: Healthy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- CARDIOSPACE II (Experimental): Test of the different devices integrated in cardiospace II.
  Interventions: Device: Test of the different devices integrated in cardiospace II

INTERVENTIONS:
Device: Test of the different devices integrated in cardiospace II — The different devices included in CARDIOSPACE II will be tested
  * Electrocardiogram
  * Vascular Doppler
  * LaserDoppler and iontophoresis
  * Brachial blood pressure
  * Continuous blood pressure recorded at the finger level
  * Ultrasound
  * Ambulatory Electrocardiogram / SAO2 (arterial oxygen saturation)

SUMMARY:
The aim of this project is to test the CARDIOSPACE II system that integrates several medical devices. This system is dedicated to physiological studies in space environment.

* Electrocardiogram
* Vascular doppler
* Laser doppler with iontophoresis
* Continuous blood pressure recording at the finger level
* Brachial blood pressure
* Ultrasound
* Ambulatory Electrocardiogram and SAO2 (arterial oxygen saturation) recorder

ELIGIBILITY:
Inclusion Criteria:

* Height between 160 et 180 cm
* Body mass index between 18 et 24
* Normal blood pressure, heart rate and cardio-pulmonary auscultation at rest
* Normal electrocardiogram
* Possibility to perform transcranial doppler
* Able to understand aims and constraints of this study
* National health insurance
* Signature of the informed consent form

Exclusion Criteria:

* Pregnant woman (Beta HCG - human chorionic gonadotropin - with urinary test) or breastfeeding
* Participating at the time to another clinical trial investigating
* Reached or surpassed the annual amount of financial compensation allowed by clinical trials (according to French regulation)
* Taking any chronic treatment
* Any sign of cardiovascular or respiration disease
* Any sign of syncopal events by questioning (>2 events per year)
* Contraindication to perform physical activity

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 4 (Actual)
Dates: Start 2021-06-28 (Actual); Primary Completion 2021-07-02 (Actual); Study Completion 2021-07-08 (Actual)

PRIMARY OUTCOMES:
Quality of the ECG signal given by CARDIOSPACE II: scale | Through study completion, an average of 6 months
  ECG signal will be estimated by investigators using a scale (from 0 to 5) 0 is a uninterpretable signal and 5 is a very clear signal without noise
Quality of the vascular Doppler signal: scale | Through study completion, an average of 6 months
  Doppler signal will be estimated by investigators using a scale (from 0 to 5) 0 is a uninterpretable signal and 5 is a very clear signal without noise
Quality of the laser doppler signal: scale | Through study completion, an average of 6 months
  Laser Doppler signal will be estimated by investigators using a scale (from 0 to 5) 0 is a uninterpretable signal and 5 is a very clear signal without noise
Quality of the ultrasound images: scale | Through study completion, an average of 6 months
  Ultrasound images will be estimated by investigators using a scale (from 0 to 5) 0 is a uninterpretable image and 5 is a very clear image
Quality of the blood pressure wave: scale | Through study completion, an average of 6 months
  Blood pressure wave signal will be estimated by by investigators using a scale (from 0 to 5) 0 is a uninterpretable signal and 5 is a very clear signal without noise
Quality of the ambulatory measurements (ECG / SAO2) | Through study completion, an average of 6 months
  ECG and SaO2 ambulatory measurements will be estimated by investigators using a scale (from 0 to 5) 0 is a uninterpretable signal and 5 is a very clear signal without noise

CONTACTS AND LOCATIONS:
Locations (1):
- CHU d'Angers, Clinical Research Center, Angers, Maine Et Loire, France